CLINICAL TRIAL: NCT03848455
Title: Multi-chip Meta-analysis of Parkinson's Disease for Clinical Validation of Small Samples of Key Genes in Disease
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Gao Xiaoya, Associate Chief Physician, Zhujiang Hospital
Other Study IDs: 2018-SJNK-008-1
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; synaptic correlation function; key gene
MeSH Terms: conditions — Parkinson Disease | interventions — Preimplantation Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — After admission, 2 tubes of venous blood (8ml) were extracted from PD group and control group respectively for genetic testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease group: 1. Patients who meet the 2016 China Parkinson's diagnostic criteria and the 2015 International Parkinson's and Movement Disorders Association (MDS) Parkinson's disease diagnostic criteria;
  2. Newly diagnosed primary PD patients, diagnosed within 3-6 months;
  3. informed consent to the study;
  4. age > 18 older.
  Interventions: Diagnostic Test: genetic diagnosis
- Non-parkinson group: Non-parkinson group inclusion criteria: age, gender-matched PD group, non-PD, non-PDS, non-neurological degenerative disease, patients without inflammatory disease and related family history; informed consent to the study; age > 18 older.
  Interventions: Diagnostic Test: genetic diagnosis

INTERVENTIONS:
Diagnostic Test: genetic diagnosis — The venous blood of the two groups of patients was taken for genetic testing, and the expression levels of PPP2CA, PPP3CB, SYNJ1, NSF and CYCS were extracted by pre-processing the genetic data of PD and non-PD patients.

SUMMARY:
The research team used meta-analytical statistical methods to integrate the results of different research groups on Parkinson's disease, using meta-analysis to find key genes related to the pathogenesis and development of Parkinson's disease, and to make small clinical results. The verification of the sample, the internal mechanism of the pathogenesis of Parkinson's disease and provide guidance and reference for subsequent experimental research.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a relatively common degenerative disease of the central nervous system. As society gradually becomes aging, the number of PD patients is increasing, but its exact pathogenesis is still not fully understood. May be related to genetic factors, environmental factors, immunological abnormalities, mitochondrial dysfunction and oxidative stress, ageing, apoptosis and other factors; the current genetic diagnosis is in the ascendant, making the understanding of the etiology and pathogenesis of Parkinson's disease more In-depth, provide more basis and means for the pathogenesis and development of Parkinson's disease, but due to the number of individual samples, operational norms and platform differences, different research groups have great differences in the results of gene chip research on Parkinson's mechanism, resulting in the reliability is poor; In order to improve the credibility of the pathogenesis of Parkinson's disease and the development of genetic diagnosis, the investigators use the statistical means of meta-analysis to integrate the results of the chip research on Parkinson's disease in different research groups and find synaptic correlation function may be closely related to the development of Parkinson's disease, PPP2CA, PPP3CB, SYNJ1, NSF, CYCS genes may be key genes in the pathogenesis of Parkinson's disease, and the expression of these genes is related to the pathogenesis and development of PD patients. the investigators will conduct a small sample validation in the clinic to explore the intrinsic mechanism of Parkinson's disease and follow-up experimental research provides guidance and reference.

ELIGIBILITY:
Inclusion Criteria:

* PD group：

  * Patients who meet the 2016 China Parkinson's diagnostic criteria and the 2015 International Parkinson's and Movement Disorders Association (MDS) Parkinson's disease diagnostic criteria
  * Newly diagnosed primary PD patients, diagnosed within 3-6 months
  * Informed consent to the study
  * Age > 18 older
* Non-PD group:

  * Age, gender-matched PD group
  * Non-PD, non-PDS, non-neurological degenerative disease, patients without inflammatory disease and related family history
  * Informed consent to the study
  * Age > 18 older

Exclusion Criteria:

* Severe craniocerebral trauma patients
* Disturbance of consciousness
* Severe organic diseases, cerebral hemorrhage, cerebral thrombosis, severe coronary heart disease and lung disease, severe liver and kidney dysfunction, severe diabetes, severe hearing And visual impairment
* History of severe brain tumors, encephalitis or brain surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From March 25, 2019 to April 25, 2019, patients with Parkinson's disease who were admitted to the Department of Neurology, Zhujiang Hospital, and healthy volunteers who recruited from population of community and students of the Southern Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoya Gao, doctor, Principal Investigator — Southern Medical University, China
Locations (1):
- Zhujiang Hospiatal, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Zhang Y, Wang Y, Xu J, Xin P, Meng Y, Wang Q, Kuang H. The Mechanisms of Traditional Chinese Medicine Underlying the Prevention and Treatment of Parkinson's Disease. Front Pharmacol. 2017 Sep 19;8:634. doi: 10.3389/fphar.2017.00634. eCollection 2017. PMID 28970800
- [Background] Lee Y, Kim MS, Lee J. Neuroprotective strategies to prevent and treat Parkinson's disease based on its pathophysiological mechanism. Arch Pharm Res. 2017 Oct;40(10):1117-1128. doi: 10.1007/s12272-017-0960-8. Epub 2017 Sep 26. PMID 28952032
- [Background] Lotankar S, Prabhavalkar KS, Bhatt LK. Biomarkers for Parkinson's Disease: Recent Advancement. Neurosci Bull. 2017 Oct;33(5):585-597. doi: 10.1007/s12264-017-0183-5. Epub 2017 Sep 21. PMID 28936761
- [Background] Walsh CJ, Hu P, Batt J, Santos CC. Microarray Meta-Analysis and Cross-Platform Normalization: Integrative Genomics for Robust Biomarker Discovery. Microarrays (Basel). 2015 Aug 21;4(3):389-406. doi: 10.3390/microarrays4030389. PMID 27600230
- [Background] Tseng GC, Ghosh D, Feingold E. Comprehensive literature review and statistical considerations for microarray meta-analysis. Nucleic Acids Res. 2012 May;40(9):3785-99. doi: 10.1093/nar/gkr1265. Epub 2012 Jan 19. PMID 22262733
- [Background] Wang X, Kang DD, Shen K, Song C, Lu S, Chang LC, Liao SG, Huo Z, Tang S, Ding Y, Kaminski N, Sibille E, Lin Y, Li J, Tseng GC. An R package suite for microarray meta-analysis in quality control, differentially expressed gene analysis and pathway enrichment detection. Bioinformatics. 2012 Oct 1;28(19):2534-6. doi: 10.1093/bioinformatics/bts485. Epub 2012 Aug 3. PMID 22863766

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Controls: healthy group inclusion criteria: age, gender-matched PD group, non-PD, non-PDS, non-neurological degenerative disease, patients without inflammatory disease and related family history; informed consent to the study; age > 18 older.
  genetic diagnosis: The venous blood of the three groups of patients was taken for genetic testing, and the expression levels of PPP2CA, PPP3CB, SYNJ1, NSF and CYCS were extracted by pre-processing the genetic data of PD and PPS patients and healthy controls .
- Parkinson's Disease Group: 1. Patients who meet the 2016 China Parkinson's diagnostic criteria and the 2015 International Parkinson's and Movement Disorders Association (MDS) Parkinson's disease diagnostic criteria;
  2. Newly diagnosed primary PD patients, diagnosed within 3-6 months;
  3. informed consent to the study;
  4. age > 18 older.
  genetic diagnosis: The venous blood of the three groups of patients was taken for genetic testing, and the expression levels of PPP2CA, PPP3CB, SYNJ1, NSF and CYCS were extracted by pre-processing the genetic data of PD ,PPS patients and healthy controls.
- Parkinson-plus Syndrome Group: 1. patients with Parkinson-plus syndrome were diagnosed according to 2017 MDS progressive supranuclear paralysis and 2017 clinical diagnostic criteria for MDS progressive supra palsy (PSP patients) and Giman standard, the 2008 American board of neurology (AAN) MSA diagnostic consensus.2.informed consent to the study; 3.age > 18 older.
  genetic diagnosis: The venous blood of the three groups of patients was taken for genetic testing, and the expression levels of PPP2CA, PPP3CB, SYNJ1, NSF and CYCS were extracted by pre-processing the genetic data of PD and PPS patients and healthy controls .
Period: Overall Study
Arm/Group | Healthy Controls | Parkinson's Disease Group | Parkinson-plus Syndrome Group
Started | 125 | 90 | 23
Completed | 125 | 90 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease Group | Healthy Controls | Parkinson-plus Syndrome Group | Total
Number analyzed (Participants) | 90 | 125 | 23 | 238
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 46 | 71 | 16 | 133
  >=65 years | 44 | 54 | 7 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.66 (11.94) | 63.42 (10.99) | 62.30 (8.13) | 63.40 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 59 | 15 | 108
  Male | 56 | 66 | 8 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 90 | 125 | 23 | 238
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 90 | 125 | 23 | 238
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 90 | 125 | 23 | 238

OUTCOME MEASURES:

1. Primary Outcome: Parkinson's Key Gene
Description: The blood of patients were taken for genetic testing and relative expression levels of the genes(These genes expression relative to a house keeping gene:GAPDH) for PPP2CA, PPP3CB, SYNJ1, NSF were extracted.The method we used is RT-PCR.
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: gene expression relative to GAPDH
Arm/Group | Parkinson's Disease Group | Healthy Controls | Parkinson-plus Syndrome Group
Number analyzed (Participants) | 90 | 125 | 23
gene expression relative to GAPDH
  PPP2CA | 1.502 [0.718 to 3.110] | 3.653 [1.990 to 5.856] | 0.916 [0.654 to 1.452]
  PPP3CB | 1.669 [0.792 to 2.947] | 2.237 [0.903 to 4.416] | 2.320 [1.110 to 3.269]
  SYNJ1 | 0.924 [0.537 to 1.585] | 4.662 [2.278 to 7.452] | 5.206 [2.541 to 6.150]
  NSF | 1.002 [0.513 to 2.150] | 3.058 [1.665 to 4.909] | 1.408 [0.864 to 2.689]
Statistical Analysis 1: Comparison: Parkinson's Disease Group vs Healthy Controls vs Parkinson-plus Syndrome Group; we use the method of RT-PCR to detect the relative expression level of PPP2CA gene in Parkinson's disease group(90 participants), healthy controls group(125 participants) and Parkinson-plus syndrome group(23 participants).This gene expression is relative to a house keeping gene GAPDH.The data were processed using 2-△△Ct. ΔCT(test) = CT(target, test) - CT(ref, test), ΔCT(calibrator) = CT(target, calibrator) - CT(ref, calibrator),ΔΔCT = ΔCT(test) - ΔCT(calibrator); Test type: Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Parkinson's Disease Group vs Healthy Controls vs Parkinson-plus Syndrome Group; we use the method of RT-PCR to detect the relative expression level of SYNJ1 gene in Parkinson's disease group(90 participants), healthy controls group(125 participants) and Parkinson-plus syndrome group(23 participants).This gene expression is relative to a house keeping gene GAPDH.The data were processed using 2-△△Ct. ΔCT(test) = CT(target, test) - CT(ref, test), ΔCT(calibrator) = CT(target, calibrator) - CT(ref, calibrator),ΔΔCT = ΔCT(test) - ΔCT(calibrator); Test type: Other; p < 0.001, Kruskal-Wallis
Statistical Analysis 3: Comparison: Parkinson's Disease Group vs Healthy Controls vs Parkinson-plus Syndrome Group; we use the method of RT-PCR to detect the relative expression level of PPP3CB gene in Parkinson's disease group(90 participants), healthy controls group(125 participants) and Parkinson-plus syndrome group(23 participants).This gene expression is relative to a house keeping gene GAPDH.The data were processed using 2-△△Ct. ΔCT(test) = CT(target, test) - CT(ref, test), ΔCT(calibrator) = CT(target, calibrator) - CT(ref, calibrator),ΔΔCT = ΔCT(test) - ΔCT(calibrator); Test type: Other; p = 0.149, Kruskal-Wallis
Statistical Analysis 4: Comparison: Parkinson's Disease Group vs Healthy Controls vs Parkinson-plus Syndrome Group; we use the method of RT-PCR to detect the relative expression level of NSF gene in Parkinson's disease group(90 participants), healthy controls group(125 participants) and Parkinson-plus syndrome group(23 participants).This gene expression is relative to a house keeping gene GAPDH.The data were processed using 2-△△Ct. ΔCT(test) = CT(target, test) - CT(ref, test), ΔCT(calibrator) = CT(target, calibrator) - CT(ref, calibrator),ΔΔCT = ΔCT(test) - ΔCT(calibrator); Test type: Other; p < 0.001, Kruskal-Wallis

2. Primary Outcome: Unified Parkinson's Disease Rating Scale 3.0（UPDRS 3.0）
Description: The total score ranges from 0 to 199( minimum score is 0 and maximum scores is 199), in which a lower score denotes a better perception of the patient's.
  Scoring the mental, behavioral and emotional, daily living activities, exercise tests, and drug treatment complications associated with UPDRS3.0 in patients with Parkinson's disease;each item 0-4 points, total score 199 points, 0-50 points: limb and body mild dysfunction, posture response normal;51-100 points: mild postural reaction disorder, self-care in daily life, loss of labor force;101-199: obvious postural reaction disorder, loss of daily life and labor force, may need help to get up and confined to wheelchair life;The more severe the symptoms of Parkinson's disease, the higher the score.
Time Frame: 2 days
Population: The "Unified Parkinson's Disease Rating Scale 3.0" is just suitable for PD patients,so there are no relative result for the group of healthy controls and Parkinson-plus syndrome group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parkinson's Disease Group: 1. Patients who meet the 2016 China Parkinson's diagnostic criteria and the 2015 International Parkinson's and Movement Disorders Association (MDS) Parkinson's disease diagnostic criteria;
  2. Newly diagnosed primary PD patients, diagnosed within 3-6 months;
  3. informed consent to the study;
  4. age > 18 older.
  genetic diagnosis: The venous blood of the two groups of patients was taken for genetic testing, and the expression levels of PPP2CA, PPP3CB, SYNJ1, NSF and CYCS were extracted by pre-processing the genetic data of PD and non-PD patients.
Arm/Group | Parkinson's Disease Group | Healthy Controls | Parkinson-plus Syndrome Group
Number analyzed (Participants) | 90 | 0 | 0
score on a scale | 61.352 (29.611) |  |

3. Primary Outcome: Non-motor Symptom Scale (NMSS)
Description: Scoring based on the patient's own situation in the last month Severity: 1 = mild; 2 = moderate; 3 = severe Frequency: 1 = very little (less than once a week); 2 = often (1 time a week); 3 = frequent (a few times a week); 4 = very frequent (every day or persist)
Time Frame: 2 days
Population: Data were not collected.
Arm/Group | Parkinson's Disease Group | Healthy Controls | Parkinson-plus Syndrome Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 years
Description: There is no Serious Adverse Events occured
Arm/Group | Parkinson's Disease Group | Healthy Controls | Parkinson-plus Syndrome Group
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/125 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/125 | 0/23
Other Adverse Events (participants affected / at risk) | 0/90 | 0/125 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT03848455/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT03848455/ICF_001.pdf